CLINICAL TRIAL: NCT05733351
Title: Multiple-Arm Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of XmAb20717 in Combination With Standard of Care Treatment in Patients With Metastatic Castration Sensitive Prostate Cancer
Brief Title: Vudalimab (XmAb20717) in Combination With Standard of Care Treatment in Patients With Metastatic Castration Sensitive Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: To review the safety data.
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Xencor, Inc. (Industry)
Responsible Party: Principal Investigator, Bassel Nazha, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004688; NCI-2023-00171 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00004688 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP5741-22 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Castration-Sensitive Prostate Carcinoma; Metastatic Prostate Adenocarcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone; Specimen Handling; Docetaxel; enzalutamide; Magnetic Resonance Spectroscopy; Glutamate Carboxypeptidase II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A (Vudalimab, Abiraterone) (Experimental): Patients receive vudalimab IV on days 1 and 15 plus abiraterone PO QD of 4-week cycles on study. Patients also undergo PSMA PET and FDG PET scans during screening. Patients also undergo CT and/or MRI scans, bone scans, and blood sample collection throughout the study.
  Interventions: Drug: Abiraterone; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: FDG-Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Procedure: PSMA PET Scan; Drug: Vudalimab
- Cohort B (Vudalimab, Enzalutamide) (Experimental): Patients receive vudalimab IV on days 1 and 15 plus enzalutamide PO QD of 4-week cycles on study. Patients also undergo PSMA PET and FDG PET scans during screening. Patients also undergo CT and/or MRI scans, bone scans, and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Enzalutamide; Procedure: FDG-Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Procedure: PSMA PET Scan; Drug: Vudalimab
- Cohort C (Vudalimab, Docetaxel, Abiraterone) (Experimental): Patients receive vudalimab IV on days 1 and 15, docetaxel IV on days 1 and 22 plus abiraterone PO QD of 6-week cycles on study. Patients also undergo PSMA PET and FDG PET scans during screening. Patients also undergo CT and/or MRI scans, bone scans, and blood sample collection throughout the study.
  Interventions: Drug: Abiraterone; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Docetaxel; Procedure: FDG-Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Procedure: PSMA PET Scan; Drug: Vudalimab

INTERVENTIONS:
Drug: Abiraterone — Given PO
  Other Names: CB 7598
  Arms: Cohort A (Vudalimab, Abiraterone); Cohort C (Vudalimab, Docetaxel, Abiraterone)
Procedure: Biospecimen Collection — Undergo blood and stool sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Cohort C (Vudalimab, Docetaxel, Abiraterone)
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi
  Arms: Cohort B (Vudalimab, Enzalutamide)
Procedure: FDG-Positron Emission Tomography — Undergo FDG PET
  Other Names: FDG; FDG-PET; FDG-PET Imaging
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: PSMA PET Scan — Undergo PSMA PET
  Other Names: Prostate-specific Membrane Antigen PET; PSMA PET
Drug: Vudalimab — Given IV
  Other Names: Anti-PD-1/Anti-CTLA-4 XmAb20717; Anti-PD1/CTLA4 Bispecific Antibody XmAb20717; PD-1 x CTLA-4 Bispecific Antibody XmAb20717; PD-1 x CTLA-4 Dual Checkpoint Inhibitor XmAb20717; XmAb 20717; XmAb20717

SUMMARY:
This phase I trial tests the safety and effectiveness of vudalimab (XmAb20717) in combination with standard of care treatment abiraterone, enzalutamide, or abiraterone plus docetaxel in treating patients with castration sensitive prostate cancer that has spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as vudalimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Adding vudalimab to standard of care treatments may be effective in treating metastatic castration sensitive prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability of vudalimab (XmAb20717) in combination with standard of care treatment in subjects with metastatic castration sensitive prostate cancer (mCSPC) as assessed by frequency and intensity of adverse events.

SECONDARY OBJECTIVE:

I. To assess the preliminary antitumor activity of vudalimab (XmAb20717) with standard of care treatment.

TERTIARY/EXPLORATORY OBJECTIVE:

I. To identify factors that may be indicative of response to vudalimab (XmAb20717) in combination with standard of care treatments.

OUTLINE: Patients are assigned to 1 of 3 cohorts.

COHORT A: Patients receive vudalimab intravenously (IV) on days 1 and 15 plus abiraterone orally (PO) once daily (QD) of 4-week cycles on study. Patients also undergo prostate-specific membrane antigen (PSMA) positron emission tomography (PET) and fludeoxyglucose (FDG) PET scans during screening. Patients also undergo computed tomography (CT) and/or magnetic resonance imaging (MRI) scans, bone scans, and blood sample collection throughout the study.

COHORT B: Patients receive vudalimab IV on days 1 and 15 plus enzalutamide PO QD of 4-week cycles on study. Patients also undergo PSMA PET and FDG PET scans during screening. Patients also undergo CT and/or MRI scans, bone scans, and blood sample collection throughout the study.

COHORT C: Patients receive vudalimab IV on days 1 and 15, docetaxel IV on days 1 and 22 plus abiraterone PO QD of 6-week cycles on study. Patients also undergo PSMA PET and FDG PET scans during screening. Patients also undergo CT and/or MRI scans, bone scans, and blood sample collection throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histologically confirmed adenocarcinoma of the prostate with metastatic disease
* Castration-sensitive status: either not have been treated with androgen deprivation therapy (ADT) (hormone therapy) or not on ADT at the time of progression

  * Participants can have received up to 3 months of ADT with luteinizing hormone-releasing hormone (LHRH) agonists or antagonists or orchiectomy with or without concurrent first-generation antiandrogens prior to enrollment, with no radiographic evidence of disease progression or rising prostate-specific antigen (PSA) prior to enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy > 12 weeks as determined by the investigator
* Hemoglobin >= 9.0 g/dl (within 28 days of cycle 1 day 1) (no transfusions allowed within 7 days of Cycle 1 Day 1 to meet entry criteria)
* White blood cell (WBC) >= 2000/uL (within 28 days of cycle 1 day 1) (after at least 7 days without growth factor support or transfusion)
* Absolute neutrophil count (ANC) >= 1,500/mcL (within 28 days of cycle 1 day 1) (after at least 7 days without growth factor support or transfusion)
* Platelets >= 100,000/mcL (within 28 days of cycle 1 day 1) (no transfusions allowed within 7 days of cycle 1 day 1 to meet entry criteria)
* Prothrombin time (PT)/ partial thromboplastin time (PTT) =< 1.5 x upper limit of normal (ULN) (within 28 days of cycle 1 day 1)
* Total bilirubin =< 1.5 institutional upper limit of normal (ULN) (within 28 days of cycle 1 day 1)
* Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) =< 3 institutional upper limit of normal (ULN) (within 28 days of cycle 1 day 1)
* Serum creatinine =< 2 mg/dL (or glomerular filtration rate >= 40 mL/min) (within 28 days of cycle 1 day 1)
* Willingness to provide pre- and post-treatment fresh tumor biopsies, if safe and medically feasible
* Male subjects must be surgically sterile or must agree to use adequate method of contraception from the time of consent until at least 120 days after the last dose of Xmab27017
* Willingness and ability of the subject to comply with scheduled visits, drug administration plan, protocol specified laboratory tests, other study procedures, and study restrictions
* Completion of all previous surgery, radiotherapy, chemotherapy, immunotherapy, or investigational therapy for the treatment of cancer >= 2 weeks before the start of study therapy. (No radiotherapy to Xmab27017 injection site within 4 weeks)
* Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier (i.e., have residual toxicities > grade 1)
* Patients who are receiving any other investigational agents or an investigational device within 21 days before administration of first dose of study drugs
* Prior treatment with any CTLA4, PD1, or PDL1, or directed immunotherapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to (investigational new drug [IND] agent[s]) or other agents used in study
* Have known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are radiologically stable, ie, are without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), are clinically stable, and are without requirement of steroid treatment for at least 14 days prior to first dose of study treatment
* Active known or suspected autoimmune disease (except that subjects are permitted to enroll if they have vitiligo; type 1 diabetes mellitus or residual hypothyroidism due to an autoimmune condition that is treatable with hormone replacement therapy only; psoriasis, atopic dermatitis, or another autoimmune skin condition that is managed without systemic therapy; or arthritis that is managed without systemic therapy beyond oral acetaminophen and nonsteroidal anti-inflammatory drugs)
* Has any condition requiring systemic treatment with corticosteroids, prednisone equivalents, or other immunosuppressive medications within 14 days prior to first dose of study drug (except that inhaled or topical corticosteroids or brief courses of corticosteroids given for prophylaxis of contrast dye allergic response are permitted.)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receipt of an organ allograft
* Known history of left ventricular ejection fraction =< 40%
* Receipt of a live-virus vaccine within 30 days prior to first dose of study drug (seasonal flu vaccines that do not contain live virus are permitted. COVID-19 vaccines are permitted)
* Known human immunodeficiency virus (HIV) positive subject with CD4+ T-cell (CD4+) counts < 350 cells/uL, or an HIV viral load greater than 400 copies/mL, or a history of an AIDS (acquired immunodeficiency syndrome)-defining opportunistic infection within the past 12 months, or who has not been on established antiretroviral therapy (ART) for at least 4 weeks prior to initiation of study drug dosing. (Effective ART is defined as a drug, dosage, and schedule associated with reduction and control of the viral load.)
* Known positive test for hepatitis C ribonucleic acid (RNA) (a subject who is hepatitis C virus [HCV] antibody positive but HCV RNA negative due to documented, curative prior antiviral treatment or natural resolution is eligible).
* Known positive test for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb; a subject whose HBsAg is negative and HBcAb is positive may be enrolled if a hepatitis B virus [HBV] deoxyribonucleic acid (DNA) test is negative, and the subject is retested for HBsAg and HBV DNA every 2 months)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Up to 70 days post treatment
  Will be assessed using the National Cancer Institute, Common Terminology Criteria for Adverse Events, Version 5.0 where, Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental activities of daily living.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to adverse event. Descriptive statistics will be used to summarize the toxicity profile of the intervention. Toxicities will be tabulated by grade, association, and cycle number.
Radiographic Progression-Free Survival | Up to 3 years
  Will be assessed per Prostate Cancer Working Group modified Response Evaluation Criteria in Solid Tumors (RECIST 1.1) as outlined in Prostate Cancer Working Group 31 (soft tissue to be assessed by RECIST 1.1, and bone disease to be assessed by Prostate Cancer Working Group 3) by radiologic evaluation.
  PSA response rate: PSA decline greater than or equal to 50% from baseline up to 24 weeks from treatment initiation.

SECONDARY OUTCOMES:
Objective Response Rate | Up to 3 years
  Will be summarized with the 2-sided 95% CI using the Clopper-Pearson method. Kaplan-Meier methods will be used to estimate median survival time or time-specific survival rate with a 95% confidence interval for rPFS or a time-to-event outcome.
PSA Response Rate | Baseline up to 24 weeks from treatment initiation
  PSA decline >= 50% and will be calculated along with 95% exact confidence intervals.
  The fold change of the numbers of CD8 T-cells or other tumor-specific T-cells before and after treatment will be described by summary statistics (mean, median, Q1, Q3, standard deviation).
PSA undetectable rate | Baseline up to 24 weeks from treatment initiation
  PSA undetectable rate will be assessed by PSA < 0.2 ng/mL up to 24 weeks from treatment initiation. Will be estimated with the Kaplan-Meier method with time-specific rate estimated with 95%CI.
Duration of response | Up to 3 years
  Will be assessed per PCWG-modified RECIST 1.1 and calculated along with 95% exact confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Bassel Nazha, MD, MPH, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT05733351/Prot_SAP_000.pdf
  • Informed Consent Form (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT05733351/ICF_001.pdf